CLINICAL TRIAL: NCT04461392
Title: Role of Myocardial Work in the Prediction of Cardiac Dysfunction and Response After Revalidation in Patients With Cancer Undergoing Chemotherapy and/or Radiotherapy
Brief Title: Exercise Response After Revalidation in Cancer Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Bernard Cosyns, Head of Department, Universitair Ziekenhuis Brussel
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BC032020_1
Record Dates: First submitted 2020-03-20; First posted 2020-07-08 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: Oncology; Cardiac Toxicity
Keywords: Echocardiography; Revalidation; Cardiovascular magnetic resonance imaging; Oncology; Radiotherapy; Chemotherapy; Cardiorespiratory exercise test
MeSH Terms: conditions — Neoplasms; Cardiotoxicity | interventions — Echocardiography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Oncology patients (Experimental): Patients diagnosed with cancer and treated with chemotherapy and/or radiotherapy
  Interventions: Diagnostic Test: Cardiorespiratory exercise test

INTERVENTIONS:
Diagnostic Test: Cardiorespiratory exercise test — * Cardiorespiratory exercise test to evaluate the exercise tolerance
  * Cardiac imaging for the assessment of the left atrium anatomy and function.
  Other Names: cardiac computed tomography; cardiac magnetic resonance; echocardiography

SUMMARY:
This study regarding oncological patients for rehabilitation after specific cancer therapy involves three aims: (1) to evaluate the predictive value of myocardial work parameters on the improvement of exercise performance after rehabilitation, (2) to determine which echocardiographic parameters are more suitable in predicting cardiac dysfunction, and (3) to evaluate the correlation between echocardiographic parameters and fibrosis detected by cardiac magnetic resonance imaging (CMR).

DETAILED DESCRIPTION:
Myocardial work (MW) provides an estimation of cardiac function by combining global longitudinal strain (GLS) with blood pressure values obtained non-invasively, being less load dependent than standard GLS. The investigator hypothesize that myocardial work could be a useful marker for predicting the exercise performance after chemotherapy and/or radiotherapy in oncological patients undergoing rehabilitation. Moreover, this study may provide additional information in optimal selection for rehabilitation programs.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with cancer
2. Undergoing chemotherapy and/or radiotherapy/hormone therapy
3. Age older than 18 years old - maximum age of 90 years old
4. Willing to enter revalidation in Universitair Ziekenhuis Brussel
5. Signed consent form

Exclusion Criteria:

1. Severe aortic stenosis defined as aortic valve aria under 0.6 cm2/m2
2. Supraventricular arrhythmias
3. Poor image quality for 2D and 3D echocardiography defined as the impossibility to examine of more than 2 adjacent segments
4. Resistant hypertension defined as uncontrolled blood pressure values under current European guidelines, Systolic Blood Pressure more than 140 mmHg and/or Diastolic Blood Pressure more than 80 mmHg
5. Lung cancer

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 191 (Estimated)
Dates: Start 2020-08 (Estimated); Primary Completion 2021-07 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Change in peak volume oxygen - VO2 (L/min) | change from baseline (before rehabilitation) at 15 months (after rehabilitation)
  represents the maximum oxygen consumption during incremental exercise that is measured during Cardiopulmonary Exercise test (CPET), being a measure of aerobic capacity of the subject
Change in the minute ventilation/carbon dioxide production (VE/VCO2) slope | change from baseline (before rehabilitation) at 15 months (after rehabilitation)
  this parameter shows the increase in ventilation in response to CO2 production, thus it measures the ventilatory efficiency
Change in the respiratory exchange ratio (RER) | change from baseline (before rehabilitation) at 15 months (after rehabilitation)
  represents the ratio between exhaled CO2 and inhale O2 may quantify the grade of the effort

SECONDARY OUTCOMES:
Change in myocardial work (MW) | change from baseline (before rehabilitation) at 15 months (after rehabilitation)
  Myocardial work (MW) is a non-invasive, less load-dependent echocardiographic parameter obtained during standard transthoracic echography using the pressure-strain loop data.
  This parameter consists of the following measurements: Global constructive work (GCW) Global wasted work (GWW), Global work index (GWI), and Global work efficiency (GWE)
Change in health status | change from baseline (before rehabilitation) at 15 months (after rehabilitation)
  Self-assessment of the generic health status using the EQ-5D-5L questionnaire. This questionnaire assesses health status in terms of five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, on a five-level scale.
  In the evaluation part, the respondents evaluate their overall health status using the visual analogue scale (EQ-VAS) from 0 ('the worst health you can imagine') - 100 ('the best health you can imagine')
Major adverse cardiovascular events (MACE) | through study completion, an average of 1 year
  nonfatal stroke, nonfatal myocardial infarction, and cardiovascular death

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Cosyns, Professor, Principal Investigator — Universitair Ziekenhuis Brussel
Locations (1):
- Universitair Ziekenhuis Brussel, Jette, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zamorano JL, Lancellotti P, Rodriguez Munoz D, Aboyans V, Asteggiano R, Galderisi M, Habib G, Lenihan DJ, Lip GYH, Lyon AR, Lopez Fernandez T, Mohty D, Piepoli MF, Tamargo J, Torbicki A, Suter TM; ESC Scientific Document Group. 2016 ESC Position Paper on cancer treatments and cardiovascular toxicity developed under the auspices of the ESC Committee for Practice Guidelines: The Task Force for cancer treatments and cardiovascular toxicity of the European Society of Cardiology (ESC). Eur Heart J. 2016 Sep 21;37(36):2768-2801. doi: 10.1093/eurheartj/ehw211. Epub 2016 Aug 26. No abstract available. PMID 27567406
- [Background] Ferreira de Souza T, Quinaglia A C Silva T, Osorio Costa F, Shah R, Neilan TG, Velloso L, Nadruz W, Brenelli F, Sposito AC, Matos-Souza JR, Cendes F, Coelho OR, Jerosch-Herold M, Coelho-Filho OR. Anthracycline Therapy Is Associated With Cardiomyocyte Atrophy and Preclinical Manifestations of Heart Disease. JACC Cardiovasc Imaging. 2018 Aug;11(8):1045-1055. doi: 10.1016/j.jcmg.2018.05.012. PMID 30092965
- [Background] Piepoli MF, Abreu A, Albus C, Ambrosetti M, Brotons C, Catapano AL, Corra U, Cosyns B, Deaton C, Graham I, Hoes A, Lochen ML, Matrone B, Redon J, Sattar N, Smulders Y, Tiberi M. Update on cardiovascular prevention in clinical practice: A position paper of the European Association of Preventive Cardiology of the European Society of Cardiology. Eur J Prev Cardiol. 2020 Jan;27(2):181-205. doi: 10.1177/2047487319893035. Epub 2019 Dec 12. PMID 31826679
- [Background] Kosmas CE, Silverio D, Sourlas A, Montan PD, Guzman E. Role of spironolactone in the treatment of heart failure with preserved ejection fraction. Ann Transl Med. 2018 Dec;6(23):461. doi: 10.21037/atm.2018.11.16. PMID 30603649
- [Background] Schrub F, Schnell F, Donal E, Galli E. Myocardial work is a predictor of exercise tolerance in patients with dilated cardiomyopathy and left ventricular dyssynchrony. Int J Cardiovasc Imaging. 2020 Jan;36(1):45-53. doi: 10.1007/s10554-019-01689-4. Epub 2019 Sep 12. PMID 31515694
- [Background] Galli E, Vitel E, Schnell F, Le Rolle V, Hubert A, Lederlin M, Donal E. Myocardial constructive work is impaired in hypertrophic cardiomyopathy and predicts left ventricular fibrosis. Echocardiography. 2019 Jan;36(1):74-82. doi: 10.1111/echo.14210. Epub 2018 Nov 29. PMID 30488501
- [Background] Ponikowski P, Voors AA, Anker SD, Bueno H, Cleland JGF, Coats AJS, Falk V, Gonzalez-Juanatey JR, Harjola VP, Jankowska EA, Jessup M, Linde C, Nihoyannopoulos P, Parissis JT, Pieske B, Riley JP, Rosano GMC, Ruilope LM, Ruschitzka F, Rutten FH, van der Meer P; ESC Scientific Document Group. 2016 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure: The Task Force for the diagnosis and treatment of acute and chronic heart failure of the European Society of Cardiology (ESC)Developed with the special contribution of the Heart Failure Association (HFA) of the ESC. Eur Heart J. 2016 Jul 14;37(27):2129-2200. doi: 10.1093/eurheartj/ehw128. Epub 2016 May 20. No abstract available. PMID 27206819
- [Background] Moneghetti KJ, Kobayashi Y, Christle JW, Ariyama M, Vrtovec B, Kouznetsova T, Wilson A, Ashley E, Wheeler MT, Myers J, Haddad F. Contractile reserve and cardiopulmonary exercise parameters in patients with dilated cardiomyopathy, the two dimensions of exercise testing. Echocardiography. 2017 Aug;34(8):1179-1186. doi: 10.1111/echo.13623. Epub 2017 Jul 6. PMID 28681553